CLINICAL TRIAL: NCT05606861
Title: Effect of Mindfulness Based Stres Reduction Intervention on Psychological Resilience of Child Nurses: Randomized Controlled Trial
Brief Title: Mindfulness Based Interventions in Pediatric Nurses
Acronym: PRoNMBSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Tülün Liman, Principal investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 69631334-300
Record Dates: First submitted 2022-10-25; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Behavior, Health
Keywords: Pediatric Nurse; Psychological Resilience; Mindfulness
MeSH Terms: conditions — Health Behavior | interventions — Nurses, Pediatric

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Mindfulness Based Intervention in pediatric nurses components was applied to this group.
  Interventions: Other: Mindfulness Based Interventions in Pediatric Nurses
- Control group (No Intervention): No procedure was conducted the control group.

INTERVENTIONS:
Other: Mindfulness Based Interventions in Pediatric Nurses — This intervention are structured mindfulness program including meditation and breathing techniques .
  Arms: Intervention group

SUMMARY:
The aim of the study was to evaluate the effect of the Mindfulness Stress Reduction Intervention on increasing the psychological resilience of pediatric nurses.

Design: This is a single-center, single-blind, randomized controlled trial

Method:

In the study, the group in which the Mindfulness-Based Stress Reduction Initiative was applied was taken as the experimental (n: 15), the unstructured group (n: 14) in which the stressful life experiences were shared as the control group. Due to the limited number of the research population (N:56), 29 nurses who agreed to participate in the study and met the inclusion criteria were included in the study without using the sampling method. This research was conducted with pediatric nurses working in the inpatient units of a children's hospital affiliated to a university in Izmir. Stress reduction training based on mindfulness, including meditation and breathing techniques, was given to the experimental group for 5 weeks. No intervention was applied to the control group.

The primary outcomes of the study were measured using the Perceived Stress Scale, the Self-Compassion Scale, the Interpersonal Reactivity Index, and Psychological Resilience Scale for Adults.

This study is important because it is the first randomized controlled study on the effect of Mindfulness Based Stress Reduction (MBSR) on resilience in nurses in our country.

In addition, the results will contribute to preventing nurses from leaving the profession in the early period, providing more flexibility and therefore safe patient care to the nursing workforce, especially in today's health system where there is a heavy nursing shortage.

ELIGIBILITY:
Inclusion Criteria:

* Working for at least one year in the children's ward,
* Older than 18 years of age,
* The working program must be suitable for the experiment schedule.

Exclusion Criteria:

* Clinical diagnosis for a psychiatric disorder,
* Long experience of meditation or yoga.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Level | For 9 weeks
  Perceived Stress Scale:The lowest score which can be obtained on the scale is 0, and the highest is 56.Higher total score means higher perceived stress level.
Psychological Resilience Level | For 9 weeks
  Psychological Resilience Scale for Adults: The minimum score on the scale is 33, and the maximum is 165. A low score on the scale indicates that the person's psychological resilience level is inadequate.
Empathy Level | For 9 weeks
  Interpersonal Reactivity Index: The scale measures different aspects of empathy. For example, the perspective-taking dimension expresses better interpersonal functioning and higher self-esteem, while the empathetic thinking dimension expresses a consistent relationship with social competence or self-esteem.
Self Compassion Level | For 9 weeks
  The Self-Compassion Scale consists of 26 Likert type items and six sub-dimensions.A higher total score on the scale indicates a higher level of self-compassion perceived by the participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No